CLINICAL TRIAL: NCT02666443
Title: Low Dose Dexamethasone as an Adjuvant to Supraclavicular Brachial Plexus Blocks: A Prospective Randomized, Double Blinded, Control Study
Brief Title: Low Dose Dexamethasone in Supraclavicular Blocks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Nathan Brown, Staff Anesthesiologist, Calgary Department of Anesthesia, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB13-1350
Record Dates: First submitted 2016-01-24; First posted 2016-01-28 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Nerve Entrapment; Ligament Injury
Keywords: brachial plexus; supraclavicular; duration; dexamethasone; block
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Nerve Compression Syndromes; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (C) (Placebo Comparator): Control intervention (no dexamethasone)
  Interventions: Drug: Control intervention (no dexamethasone)
- Peri-neural (N) (Experimental): Peri-neural Dexamethasone 1 mg
  Interventions: Drug: Peri-neural Dexamethasone 1 mg
- Intravenous (Experimental): Intravenous Dexamethasone 1 mg
  Interventions: Drug: Intravenous Dexamethasone 1 mg

INTERVENTIONS:
Drug: Control intervention (no dexamethasone) — Patients receive a supraclavicular brachial plexus block with 30 mL of solution containing 0.5% bupivacaine, 1:400,000 epinephrine, 0.1 mL normal saline, and an intravenous solution of 50 mL normal saline.
  Other Names: Control
  Arms: Control (C)
Drug: Peri-neural Dexamethasone 1 mg — Patients receive a supraclavicular brachial plexus block with 30 mL of solution containing 0.5% bupivacaine, 1:400,000 epinephrine, 0.1 mL dexamethasone 1% (1 mg dexamethasone), and an intravenous solution of 50 mL normal saline.
  Other Names: Peri-neural
  Arms: Peri-neural (N)
Drug: Intravenous Dexamethasone 1 mg — Patients receive a supraclavicular brachial plexus block with 30 mL of solution containing 0.5% bupivacaine, 1:400,000 epinephrine, 0.1 mL normal saline, and an intravenous solution of 49.9 mL normal saline with 0.1mL dexamethasone 1%
  Other Names: IV
  Arms: Intravenous

SUMMARY:
Brachial plexus nerve blocks provide superior analgesia over opioids while avoiding unwanted side effects. Single shot blocks with local anesthetic alone usually do not last the duration of the acute post-surgical pain period. This has led to the exploration of multiple adjuvants to increase the duration of single shot blocks, the most promising adjuvant being dexamethasone.

Peri-neural administration is an off-label use of dexamethasone. While no adverse events have been reported in human clinical studies, logic would dictate that we minimize the dose needed to produce the desired effect. Most studies thus far have used peri-neural dexamethasone doses ranging from 4-10 mg. However, Albrecht et al. found no difference in block duration comparing 4 mg and 8 mg doses while Liu et al. reported equivalent block duration using doses of 1, 2 and 4 mg.

Recent studies have evaluated whether systemic and peri-neural administrations of dexamethasone are equivalent, which would in turn imply a site of action. Results have been mixed. Four studies concluded peri-neural and intravenous administration are equivalent at prolonging analgesia, though one study had methodological errors, including the administration of intravenous dexamethasone to all patients. All of these studies used dexamethasone doses of 8 to 10 mg. One study where a lower dose (4 mg) was used found that peri-neural administration prolonged block duration whereas intravenous did not.

With that, the rationale of our study is to determine if equivalent block-prolonging analgesia can be achieved using low dose (1 mg) dexamethasone given peri-neural or intravenous. Clinical experience at our centre has been that 1 mg dexamethasone added to 20 mL produces similar block duration to that reported in published studies using higher doses.

DETAILED DESCRIPTION:
The investigators will evaluate the block-prolonging efficacy of dexamethasone 1 mg in supraclavicular blocks. The investigators will be answering essentially two questions. First, how long do supraclavicular blocks last when low dose dexamethasone is used as an adjunct. Only one study has looked at doses this low (Liu et al. 2015). Some methodological problems with this study include evaluation of shoulder surgery using supraclavicular blocks, which may or may not cover the posterior port site; use of the endpoint of "time to first analgesic", which may or may not indicate actual block duration; and low numbers powered to 80%, which may yield spurious results. To avoid these issues the investigators chose upper limb surgery, a type of block which will definitely cover the entire surgical site, and an endpoint of time to first pain at surgical site, regardless of whether analgesic is needed. The investigators are also powering to 95% and recruiting higher numbers of patients.

The second question evaluates the efficacy of 1 mg of intravenous dexamethasone. The study is powered to address this question, but in doing so is also powered adequately to address the first question. Studies to date have mixed results and methodological errors. No other studies have evaluated this dose of intravenous dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 - 80 years
* BMI equal to or less than 35
* Upper limb surgery
* Normal pre-operative sensation in the operative limb

Exclusion Criteria:

* Pre-operative opioid greater than 4 Tylenol #3 per day (or equivalent)
* Pre-existing, fluctuating neurologic injury involving operative upper limb
* Patient refusal or patient inability to provide consent
* Suspected inability to comply with study procedures, including language difficulties or medical history and/or concomitant disease (skin infection at site of needle insertion) as judged by the investigator or attending anesthesiologist, reason for exclusion will be recorded.
* Patient pregnancy
* Patient BMI > 35
* Patient allergy to any of the drugs used in the protocol
* Surgical concern of postoperative neurological injury from surgical manipulation.
* Brittle diabetics
* Other contraindication to receiving a block (coagulopathy, significant respiratory risk, etc.)
* Surgeon refusal (e.g. concerns about compartment syndrome); reason for exclusion will be recorded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Time to first sensation of pain at the surgical site. | 72 hours

SECONDARY OUTCOMES:
duration of motor blockade | 72 hours
  time (in hours) to return of full pre-operative strength in the operative limb
morphine or morphine equivalent usage in the first 48 h postoperatively | 48 hours
incidence of nausea and vomiting and pruritus in the first 48 h | 48 hours
numerical rating scale (NRS) pain scores at 8 h, 24 h, 48 h, and post-operative day 7 | 7 days
residual paraesthesias or motor blockade at 7 days. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Nathan JD Brown, BMSc, MD, Principal Investigator — University of Calgary
Locations (1):
- South Health Campus, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
I am not sure what the entirety of a "yes" answer entails, or with whom the data would be shared. Hence, undecided.

REFERENCES:
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394
- [Background] Noss CD, MacKenzie LD, Kostash MA. Adjuvant dexamethasone: innovation, farce, or folly? Reg Anesth Pain Med. 2014 Nov-Dec;39(6):540-5. doi: 10.1097/AAP.0000000000000148. No abstract available. PMID 25275574
- [Background] Choi S, Rodseth R, McCartney CJ. Effects of dexamethasone as a local anaesthetic adjuvant for brachial plexus block: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2014 Mar;112(3):427-39. doi: 10.1093/bja/aet417. Epub 2014 Jan 10. PMID 24413428
- [Background] Huynh TM, Marret E, Bonnet F. Combination of dexamethasone and local anaesthetic solution in peripheral nerve blocks: A meta-analysis of randomised controlled trials. Eur J Anaesthesiol. 2015 Nov;32(11):751-8. doi: 10.1097/EJA.0000000000000248. PMID 25774458
- [Background] Albrecht E, Kern C, Kirkham KR. A systematic review and meta-analysis of perineural dexamethasone for peripheral nerve blocks. Anaesthesia. 2015 Jan;70(1):71-83. doi: 10.1111/anae.12823. Epub 2014 Aug 14. PMID 25123271
- [Background] Knight JB, Schott NJ, Kentor ML, Williams BA. Neurotoxicity of common peripheral nerve block adjuvants. Curr Opin Anaesthesiol. 2015 Oct;28(5):598-604. doi: 10.1097/ACO.0000000000000222. PMID 26207854
- [Background] Williams BA, Hough KA, Tsui BY, Ibinson JW, Gold MS, Gebhart GF. Neurotoxicity of adjuvants used in perineural anesthesia and analgesia in comparison with ropivacaine. Reg Anesth Pain Med. 2011 May-Jun;36(3):225-30. doi: 10.1097/AAP.0b013e3182176f70. PMID 21519308
- [Background] Williams BA, Butt MT, Zeller JR, Coffee S, Pippi MA. Multimodal perineural analgesia with combined bupivacaine-clonidine-buprenorphine-dexamethasone: safe in vivo and chemically compatible in solution. Pain Med. 2015 Jan;16(1):186-98. doi: 10.1111/pme.12592. Epub 2014 Oct 23. PMID 25339320
- [Background] Castillo J, Curley J, Hotz J, Uezono M, Tigner J, Chasin M, Wilder R, Langer R, Berde C. Glucocorticoids prolong rat sciatic nerve blockade in vivo from bupivacaine microspheres. Anesthesiology. 1996 Nov;85(5):1157-66. doi: 10.1097/00000542-199611000-00025. PMID 8916834
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Waldron NH, Jones CA, Gan TJ, Allen TK, Habib AS. Impact of perioperative dexamethasone on postoperative analgesia and side-effects: systematic review and meta-analysis. Br J Anaesth. 2013 Feb;110(2):191-200. doi: 10.1093/bja/aes431. Epub 2012 Dec 5. PMID 23220857
- [Background] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Background] Rahangdale R, Kendall MC, McCarthy RJ, Tureanu L, Doty R Jr, Weingart A, De Oliveira GS Jr. The effects of perineural versus intravenous dexamethasone on sciatic nerve blockade outcomes: a randomized, double-blind, placebo-controlled study. Anesth Analg. 2014 May;118(5):1113-9. doi: 10.1213/ANE.0000000000000137. PMID 24686045
- [Background] Fredrickson Fanzca MJ, Danesh-Clough TK, White R. Adjuvant dexamethasone for bupivacaine sciatic and ankle blocks: results from 2 randomized placebo-controlled trials. Reg Anesth Pain Med. 2013 Jul-Aug;38(4):300-7. doi: 10.1097/AAP.0b013e318292c121. PMID 23698496
- [Background] Abdallah FW, Johnson J, Chan V, Murgatroyd H, Ghafari M, Ami N, Jin R, Brull R. Intravenous dexamethasone and perineural dexamethasone similarly prolong the duration of analgesia after supraclavicular brachial plexus block: a randomized, triple-arm, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2015 Mar-Apr;40(2):125-32. doi: 10.1097/AAP.0000000000000210. PMID 25629321
- [Background] Kawanishi R, Yamamoto K, Tobetto Y, Nomura K, Kato M, Go R, Tsutsumi YM, Tanaka K, Takeda Y. Perineural but not systemic low-dose dexamethasone prolongs the duration of interscalene block with ropivacaine: a prospective randomized trial. Local Reg Anesth. 2014 Apr 5;7:5-9. doi: 10.2147/LRA.S59158. eCollection 2014. PMID 24817819
- [Background] Liu J, Richman KA, Grodofsky SR, Bhatt S, Huffman GR, Kelly JD 4th, Glaser DL, Elkassabany N. Is there a dose response of dexamethasone as adjuvant for supraclavicular brachial plexus nerve block? A prospective randomized double-blinded clinical study. J Clin Anesth. 2015 May;27(3):237-42. doi: 10.1016/j.jclinane.2014.12.004. Epub 2015 Jan 28. PMID 25637938
- [Background] Bolin ED, Wilson S. Perineural Versus Systemic Dexamethasone: Questions Remain Unanswered. Reg Anesth Pain Med. 2015 Jul-Aug;40(4):393-4. doi: 10.1097/AAP.0000000000000262. No abstract available. PMID 26079360
- [Background] Beecroft CL, Coventry DM. Anaesthesia for shoulder surgery. Continuing Education in Anaesthesia, Critical Care & Pain 2008 ; 8: 193-98
- [Background] Perlas A, Lobo G, Lo N, Brull R, Chan VW, Karkhanis R. Ultrasound-guided supraclavicular block: outcome of 510 consecutive cases. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):171-6. doi: 10.1097/AAP.0b013e31819a3f81. PMID 19282715
- [Background] Ultrasound for Regional Anesthesia, Supraclavicular Block. 2008; http://www.usra.ca/supneedle.php accessed September 22, 2015
- [Background] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Background] Shrestha BR, Maharjan SK, Shrestha S, Gautam B, Thapa C, Thapa PB, Joshi MR. Comparative study between tramadol and dexamethasone as an admixture to bupivacaine in supraclavicular brachial plexus block. JNMA J Nepal Med Assoc. 2007 Oct-Dec;46(168):158-64. PMID 18340366